CLINICAL TRIAL: NCT04146740
Title: Effects of Structured Exercise Regime for the Management of Gestational Diabetes Mellitus (GDM) - Bio Psychosocial Perspectives.
Brief Title: Effects of Structured Exercise Regime in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2019/1
Record Dates: First submitted 2019-08-26; First posted 2019-10-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Gestational Diabetes Mellitus
Keywords: exercise; pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Exercise Group (Experimental): Structured Exercise Group will receive medical and dietary interventions like insulin plus structured aerobic exercise regime of moderate intensity by using stationary cycle (3-5 MET) 10 min, brisk walk 10 min The combination of Stabilization exercise (10 repetitions) and PFM training ( 20 repetitions set).
  Relaxation therapy including Mitchells physiological relaxation technique (10 repeatitions) alongwith deep breathing exercises.
  Life style modification with postural guidance and back care would also be followed.
  Exercise dosage would be twice a week for 05 weeks while exercise duration will be 45 to 50 min session under Physio supervision and home plan of 10 min exercise daily. Total 150 min per week. Data will be recorded at baseline then after treatment of 5 weeks.
  Interventions: Other: Structured Exercise for Experimental (Structured Exercise) Group; Behavioral: Control treatment for both groups
- Control Group (Active Comparator): Control Group will receive no structured exercise regime only the group will be receiving medical and dietary interventions like insulin in addition of the postural education and back care from Physical Therapist due to ethical concerns and their outcomes will be observed at the baseline and then after 05 weeks.
  Interventions: Behavioral: Control treatment for both groups

INTERVENTIONS:
Other: Structured Exercise for Experimental (Structured Exercise) Group — Structured aerobic exercise regime of moderate intensity by using stationary cycle (3-5 MET) 10 min, brisk walk 10 min.
  The combination of Stabilization exercise (10 repeatitions) and PFM training ( 20 repeatitions set).
  Relaxation therapy including Mitchells physiological relaxation technique (10 repetitions) along with deep breathing exercises.
  Arms: Structured Exercise Group
Behavioral: Control treatment for both groups — Medical and dietary interventions like insulin in addition of the postural education and back care from Physical Therapist.

SUMMARY:
Rehabilitation in the field of Obstetrics is an emerging field worldwide although it is still very much neglected in a country like Pakistan. Increasing prevalence of GDM has highlighted the importance of rehabilitation in this specific area. In USA upto14% of pregnancies get GDM problem, 6.8 to 10.4 % in China while in India 27.5% which is exceptionally high. Similarly in Pakistan it has become a common issue.

Many observational studies have been done to find the risk factors and causes of GDM. However to the best of investigator's knowledge no experimental study have been done so far on the effects of exercise on physical, physiological and psychological aspects of GDM. Hence a randomized control trial is planned on diagnosed GDM patients in Fauji Foundation Hospital Rawalpindi who will recieve supervised structured exercise regeme for 5 weeks and their data will be recorded using reliable tools at the baseline and after 5 weeks to assess the effects of exercise.

DETAILED DESCRIPTION:
GDM is a medical condition of high maternal glucose level which is diagnosed only when women are pregnant and overcome after pregnancy. It results in various maternal and neonatal complications like caeserean delivery in mothers and obesity in children. Women having GDM have greater risk of diabetes and cardiovascular problems later in life which is threatening for us. Obese women are at increased risk of developing GDM and it is also a risk factor for developing high blood pressure and protein in the urine after 20 weeks of pregnancy that condition is known as preeclampsia.

Many studies have shown that physically active women are less prone to develop GDM as compare to those women who have sedentary life style which draws attention towards the role of antenatal exercises for prevention and management of GDM and has become the first line treatment in developed countries. In addition to obesity and sedentary life style other known risk factors are family history, age of mother and number of children but there is no definite single cause of GDM yet discovered.

Exercises programs during pregnancy are not usually practiced in our population and routine domestic activities are considered as enough for fitness. We have a common myth that pregnant women should not do treadmill or stationary cycle or any other aerobic activity which is really wrong and resulting in problems like GDM. Women following moderate exercise programs during their pregnancy have reported reduction in daily insulin administration dosage in comparison with women not doing any prescribed exercise. As Gestational weight gain is a major risk factor for GDM, exercises have given evidence to facilitate weight reduction.

Exercise programs prescribed by physical therapists during pregnancy for preventing and managing GDM are considered useful and recommended by researchers and practitioners around the world but in developing countries like Pakistan, women are not receiving this method of treatment due to lack of awareness in general public, lack of referral system from gynaecologists and obstetricians and unavailability of women health Physical therapists in hospital set ups.

This study will provide data showing the effects of exercise in biomarkers level and give the option of treatment to obstetricians.

This will fill the research gap in the area of rehabilitation in GDM. This will also highlight the importance of women health physical therapists in obstetric conditions as there is less awareness of this speciality in Pakistan.

This will provide the data regarding which type, intensity and duration of exercise should be recommendable while treating GDM.

This study will open new doors for researchers to do long term studies on different biomarkers with different exercise types.

ELIGIBILITY:
Inclusion Criteria:

1. Women with age of 20 to 40 years and gestational age more than 20 weeks.
2. Diagnosed Gestational diabetes mellitus patients
3. Must be able to do 6 min walk test and lie under severity level 6 on the 0-10 Borg scale of breathlessness -

Exclusion Criteria:

1. Diagnosed neurological and cardiopulmonary problems.

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females only.
Enrollment: 80 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
HbA1c | 5 weeks
  HbA1c will be assessed at the base line and at the end of 5 weeks session. Lower score shows better outcome.
Blood Pressure | 5 weeks
  Change in the Values of Blood pressure will be assessed at base line and at the end of 5 weeks session.
Lipid profile | 5 weeks
  Lipid profile will be assessed at the base line and at the end of 5 weeks session
Renal function test (RFT) | 5 weeks
  RFT will be assessed at the base line and at the end of 5 weeks session. Lower score shows better outcome.
C reactive protein | 5 weeks
  C reactive protein will be assessed at the base line and at the end of 5 weeks session. Lower score shows better outcome.
Heart rate | 5 weeks
  Change in the heart rate will be assessed at base line and at the end of 5 weeks session.
Respiratory rate | 5 weeks
  Change in the respiratory rate will be assessed at base line and at the end of 5 weeks.
Blood glucose level | 5 weeks
  Change in the blood glucose level will be assessed at base line and at the end of 5 weeks session.

SECONDARY OUTCOMES:
Gestational weight gain | 5 weeks
  Gestational weight gain by recording weight of women in pounds and gestational age in weeks at baseline and then after 5 weeks.
Edinburgh Post Natal Depression scale (Punjabi version) | 5 weeks
  The score of Depression using Edinburgh Post Natal Depression scale (Punjabi version). Each answer is given on a score of 0-3 . Maximum score is 30 A score of 10 or higher indicates that depressive symptoms have been

CONTACTS AND LOCATIONS:
Overall Officials: Wardah Ajaz Qazi, BS-PT, PP-DPT, PhD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aviram A, Guy L, Ashwal E, Hiersch L, Yogev Y, Hadar E. Pregnancy outcome in pregnancies complicated with gestational diabetes mellitus and late preterm birth. Diabetes Res Clin Pract. 2016 Mar;113:198-203. doi: 10.1016/j.diabres.2015.12.018. Epub 2016 Jan 12. PMID 26810272
- [Background] Wang C, Guelfi KJ, Yang HX. Exercise and its role in gestational diabetes mellitus. Chronic Dis Transl Med. 2016 Dec 20;2(4):208-214. doi: 10.1016/j.cdtm.2016.11.006. eCollection 2016 Dec. PMID 29063044
- [Background] Bain E, Crane M, Tieu J, Han S, Crowther CA, Middleton P. Diet and exercise interventions for preventing gestational diabetes mellitus. Cochrane Database Syst Rev. 2015 Apr 12;(4):CD010443. doi: 10.1002/14651858.CD010443.pub2. PMID 25864059
- [Background] Barquiel B, Herranz L, Hillman N, Burgos MA, Grande C, Tukia KM, Bartha JL, Pallardo LF. HbA1c and Gestational Weight Gain Are Factors that Influence Neonatal Outcome in Mothers with Gestational Diabetes. J Womens Health (Larchmt). 2016 Jun;25(6):579-85. doi: 10.1089/jwh.2015.5432. Epub 2016 Feb 26. PMID 26918922
- [Background] Brankica K, Valentina VN, Slagjana SK, Sasha JM. Maternal 75-g OGTT glucose levels as predictive factors for large-for-gestational age newborns in women with gestational diabetes mellitus. Arch Endocrinol Metab. 2016 Feb;60(1):36-41. doi: 10.1590/2359-3997000000126. PMID 26909480